CLINICAL TRIAL: NCT06951568
Title: Study of the Effect of Peripheral Somatosensory Stimulation on the Functionality of Patients With Cerebral Palsy and Reduced Mobility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Facultat de ciencies de la Salut Universitat Ramon Llull (Other)
Collaborators: Cerebral Palsy Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-04-09
Record Dates: First submitted 2025-04-20; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The 20 participants will be divided into two groups of 10 people. The first group (Group A) will begin the intervention with both the physiotherapy protocol and somatosensory stimulation, while the second group (Group B) will start with the physiotherapy protocol only. At the midpoint of the intervention, in week 6, the groups will switch: Group A will then receive only the physiotherapy protocol, and Group B will begin receiving somatosensory stimulation alongside the physiotherapy protocol. Both groups will continue under these conditions until week 12, marking the end of the intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Intervention INITIAL (Experimental): Group INITIAL will begin the intervention with both the physiotherapy protocol and somatosensory stimulation, At the midpoint of the intervention, in week 6, the groups will switch: Group INITIAL will then receive only the physiotherapy protocol. Both groups will continue under these conditions until week 12, which marks the end of the protocol.
  Interventions: Other: Physical Exercise Program
- Group Intervention CROSSED (Active Comparator): Group CROSSED will start with the physiotherapy protocol only. At the midpoint of the intervention, in week 6, the groups will switch: Group CROSSED will receive somatosensory stimulation alongside physiotherapy. Both groups will continue under these conditions until week 12, which marks the end of the protocol.
  Interventions: Other: Physical Exercise Program

INTERVENTIONS:
Other: Physical Exercise Program — The physiotherapy protocol has been developed using the GMFCS scale as a reference. Based on this assessment, each patient's level is determined according to their functional motor abilities, limitations, and use of assistive or mobility devices. Each protocol consists of a total of five exercises: two general exercises and three specific exercises focused on the phases of the corresponding transfer and on skills common to all transfers. Rest periods of 2 minutes and 30 seconds are provided between exercises to ensure adequate recovery and a safe progression. The somatosensory stimulation will consist of intermittent mechanical pressure applied to the skin over the neuromuscular motor points of the quadriceps and gastrocnemius muscles. T

SUMMARY:
Cerebral palsy (CP) is a permanent neurological disorder that affects movement and posture, caused by an injury to the developing brain. It may also be accompanied by cognitive, hearing, and speech impairments, as well as epilepsy. Although it is a condition that manifests in childhood, its effects persist throughout life, posing specific challenges in mobility and functionality during adulthood. Although physiotherapy is a key component in the rehabilitation of children with CP and helps adults manage pain and improve motor function, many adults with CP do not receive the treatment they need. Barriers such as financial difficulties, transportation issues, and the lack of physiotherapists specialized in CP affect both access to and the quality of care. Even when physiotherapy is provided, adults with CP are often less satisfied with the services compared to children.The aim of this study is to promote the recovery of motor function in adults with cerebral palsy through sensory stimulation of the lower limbs, as part of an intensive motor rehabilitation program. This program seeks to foster autonomy in movements and transfers, as well as active participation in daily life activities.

DETAILED DESCRIPTION:
Objective: To evaluate the impact of peripheral somatosensory stimulation on motor function in adults with cerebral palsy.

Methods: Experimental, crossover, and randomized. Each participant will serve as their own control and will be assessed under both stimulation (experimental) and non-stimulation (control) conditions.The sample will be one of convenience and will consist of the voluntary participation of 20 adults diagnosed with cerebral palsy who have reduced mobility and are institutionalized at the residence of the Catalan Foundation for Cerebral Palsy (FCPC).The physical exercise program will last for 2 days per week over a period of 12 consecutive weeks, with prior agreement from the center's management and their participation in the study. The 20 participants will be divided into two groups of 10 people. The first group (Group A) will begin the intervention with both the physiotherapy protocol and somatosensory stimulation, while the second group (Group B) will start with the physiotherapy protocol only. At the midpoint of the intervention, in week 6, the groups will switch: Group A will then receive only the physiotherapy protocol, and Group B will begin receiving somatosensory stimulation alongside the physiotherapy protocol. Both groups will continue under these conditions until week 12, marking the end of the intervention.

ELIGIBILITY:
Inclusion Criteria

* Adults with a medical diagnosis of cerebral palsy
* Age: 18-50 years
* Reduced mobility classified as levels I, II, or III according to the GMFCS
* Ability to participate in functional assessments with the support of the clinical team
* Ability to understand informed consent or have a legal representative who can provide consent on their behalf

Exclusion Criteria

* Patients with cerebral palsy who have severe cognitive impairments that hinder understanding of instructions or participation in assessments
* Adults with cerebral palsy who present with medical conditions that may interfere with the intervention, such as severe cardiovascular disease or major neurological disorders
* Individuals with cerebral palsy who are participating in another intervention study during the same period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-02 (Estimated); Primary Completion 2025-07-02 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Rivermead Mobility Index (RMI) | On the third day after the start of the intervention, in week 6, and in week 12.
  To evaluate the level of functional mobility, focusing on tasks such as turning over, walking, and climbing stairs.
  0-5 points: severely limited mobility.
  6-10 points: moderately limited mobility.
  11-15 points: mildly limited or good functional mobility.

SECONDARY OUTCOMES:
the Trunk Impairment Scale. | On the third day after the start of the intervention, in week 6, and in week 12.
  To analyze trunk postural control 0 points: complete absence of trunk control.
  1-7 points: severely impaired trunk control.
  8-15 points: moderately impaired trunk control.
  16-23 points: good trunk control (mild impairment or normal function).
number of repetitions | On the third day after the start of the intervention, in week 6, and in week 12.
  To evaluate the number of repetitions in the specific exercises of the protocol
The time taken to perform the movement | On the third day after the start of the intervention, in week 6, and in week 12.
  time required for execution and the completeness of the performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro Victor López Plaza, Barcelona, Spain